CLINICAL TRIAL: NCT06397300
Title: Comparison of Ultrasound Guided Bilateral Erector Spinae Plane Block, Ultrasound Guided Bilateral Quadratus Lumborum Block and Lumbar Epidural for Postoperative Analgesia in Patients Undergoing Total Abdominal Hysterectomy ; a Prospective Randomized Clinical Trial
Brief Title: Comparison of US Bilateral Erector Spinae Plane Block, US Bilateral Quadratus Lumborum Block and Lumbar Epidural for Postoperative Analgesia in Patients Undergoing Total Abdominal Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ahmed Mohamed Soliman, lecturer of anesthesia, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AP2312-201-095; IRB00004025 (Other: National Cancer Institute Cairo university)
Record Dates: First submitted 2024-04-18; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Comparison of US Bilateral Erector Spinae Plane Block, US Bilateral Quadratus Lumborum Block and Lumbar Epidural
Keywords: Analgesics; Opioids; Postoperative Pain; Nerve block; ultrasound; Hysterectomy; cancer; ovarian neoplasm; uterine carcinoma
MeSH Terms: conditions — Pain, Postoperative; Neoplasms; Ovarian Neoplasms | interventions — Parapsychology; Dental Occlusion

STUDY DESIGN:
Intervention Model Description: To determine the analgesic effect of US Bilateral Erector Spinae Plane Block, US Bilateral Quadratus Lumborum Block and Lumbar Epidural for Postoperative Analgesia in Patients Undergoing Total Abdominal Hysterectomy regarding the following:
  1. Post-operative opioid (morphine) consumption in the 1st 24 hours
  2. Postoperative Numeric Pain Rating Scale. 3. Effect on hemodynamics: Mean arterial blood pressure and Heart rate. 4. Intraoperative fentanyl consumption. 5. Duration of analgesic effect
Who Masked: Participant, Investigator
Masking Description: The patients will be randomly assigned into two equal comparable groups using computer- generated random numbers in opaque closed envelopes, each of which will include 30 patients. Randomization will be done by statistician and each group of the patient will revealed only when the included patient is transferred to preanesthetic room.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- bilateral Ultrasound guided erector spinae plane (ESP) block (Active Comparator): . To perform ESP block in the lateral position bilaterally, a linear transducer is placed in a longitudinal parasagittal orientation and erector spinae muscle, trapezius muscle, rhomboid major muscle and transverse process are visualized and local anesthetic is injected (0.25% bupivacaine 20 ml in each side) in the area between transverse process and erector spinae muscle at T10 level.
  Interventions: Procedure: bilateral Ultrasound guided erector spinae plane (ESP) block
- quadratus lumborum block (Active Comparator): In the lateral decubitus position. Right block will be performed; the patient will then repositioned for the left block. An ultrasound device with a convex probe (5-8 MHz) will be placed in the mid-axillary line just above the iliac crest. Then, scan dorsally to keep the transverse orientation until seeing the aponeurosis of the transverses abdominus muscle and by following this aponeurosis, QL muscle will be visualized with its attachment to the lateral edge of the transverse process of the L2 vertebral body and visualize the thoracolumbar fascia at the lateral edge of the QL muscle. A spinal needle (20G) will be inserted in-plane from the anterior to posterior direction, and the tip of the needle will be advanced anterior to the QL muscle. The target site for injection is the plane between the quadratus lumborum and psoas major muscles. This will be followed by injection of 0.25% bupivacaine 20 ml in each side.
  Interventions: Procedure: quadratus lumborum block
- lumbar epidural (Active Comparator): under strict aseptic precautions, lumbar epidural was performed for patients in Group III using a 16-gauge Touhy epidural needle by a median approach. The T12 - L1 or L1 - L2 interspaces was chosen for the injection.
  The epidural space identified by the loss of resistance technique. The catheter was advanced 4 cm cephalad. When the aspiration test results for blood and cerebrospinal fluid were negative, a test dose of (3 mL) 2% lidocaine with 1: 200,000 adrenaline was given after the placement of the epidural catheter.
  Then this will be followed by injection of 0.25% bupivacaine 15 ml as a single injection after induction of general anesthesia.
  Interventions: Procedure: lumbar epidural

INTERVENTIONS:
Procedure: bilateral Ultrasound guided erector spinae plane (ESP) block — To perform ESP block in the lateral position bilaterally ,the skin will be disinfected with 70% alchol bilaterally and a linear transducer is placed in a longitudinal parasagittal orientation and erector spinae muscle, trapezius muscle, rhomboid major muscle (rhomboid major muscle is absent below T6 level) and transverse process are visualized and local anesthetic is injected (0.25% bupivacaine 20 ml in each side) in the area between transverse process and erector spinae muscle at T10 level.
  Arms: bilateral Ultrasound guided erector spinae plane (ESP) block
Procedure: quadratus lumborum block — In the lateral decubitus position. Right block will be performed; the patient will then repositioned for the left block. An ultrasound device with a convex probe (5-8 MHz) will be placed in the mid-axillary line just above the iliac crest. Then, scan dorsally to keep the transverse orientation until seeing the aponeurosis of the transverses abdominus muscle and by following this aponeurosis, QL muscle will be visualized with its attachment to the lateral edge of the transverse process of the L2 vertebral body and visualize the thoracolumbar fascia at the lateral edge of the QL muscle. A spinal needle (20G) will be inserted in-plane from the anterior to posterior direction, and the tip of the needle will be advanced anterior to the QL muscle. The target site for injection is the plane between the quadratus lumborum and psoas major muscles. This will be followed by injection of 0.25% bupivacaine 20 ml in each side.
  Arms: quadratus lumborum block
Procedure: lumbar epidural — under strict aseptic precautions, lumbar epidural was performed for patients in Group III using a 16-gauge Touhy epidural needle by a median approach. The T12 - L1 or L1 - L2 interspaces was chosen for the injection.
  The epidural space identified by the loss of resistance technique. The catheter was advanced 4 cm cephalad. When the aspiration test results for blood and cerebrospinal fluid were negative, a test dose of (3 mL) 2% lidocaine with 1: 200,000 adrenaline was given after the placement of the epidural catheter.
  Then this will be followed by injection of 0.25% bupivacaine 15 ml as a single injection after induction of general anesthesia.
  Arms: lumbar epidural

SUMMARY:
The investigators hypothesize that US Bilateral Erector Spinae Plane Block, US Bilateral Quadratus Lumborum Block and Lumbar Epidural for Postoperative Analgesia in Patients Undergoing Total Abdominal Hysterectomy resulting in reducing myofascial pain and opioid consumption.

DETAILED DESCRIPTION:
Background and Rationale:

Gynecological cancers comprise 10-15% of women's cancers, mainly affecting women post-reproductive age but posing threats to fertility for younger patients.

The goal of postoperative pain control is to reduce the negative consequences associated with acute postsurgical pain and help the patient make a smooth transition back to normal function. Traditionally, opioid analgesic therapy has served as the mainstay of treatment for acute postoperative pain. However, the recent rise in morbidity and mortality associated with opioid misuse has led to increasing demands for more investigative efforts into developing pain treatment strategies that place more emphasis on using a multimodal approach. These efforts have proved to be challenging, as the subjective nature of pain perception further complicates the ability to achieve satisfactory pain control. Furthermore, specific patient comorbidities and social factors may predispose patients to have increased pain perception.

Approximately 75 percent of patients who undergo surgery experience acute postoperative pain, which is often medium-high in severity. Less than half of patients undergoing surgery report adequate postoperative pain relief. This percentage presents a significant problem as inadequate postoperative pain control may lead to adverse physiologic effects among patients in the immediate postoperative period and place them at increased risk of developing chronic pain associated with the procedure. Severe persistent postoperative pain affects 2 to 10 percent of adults.

Multiple peer-reviewed publications address the topic of postoperative pain control in gynecologic oncology surgery. Because many of these surgeries require large laparotomy incisions, patients frequently receive intravenous opioids for pain control. Patient-controlled analgesia, or PCAs, are often used as the mechanism of delivery as they allow patients to deliver pain medications based on their perceived needs. Intravenous opioids are associated with undesired side effects, including nausea, pruritus, hallucinations, and delay in the return of bowel function, which may ultimately lead to prolonged hospitalization and extended recovery times. The use of ultrasonographic technology in regional anesthesia practice has not only eased the application of nerve blocks and interfascial blocks but also led to the definition and practical use of many new interfascial blocks. Thoracoabdominal/thoracolumbar blocks - also named as truncal blocks, have gained popularity recently with the number of such defined blocks increasing substantially.

Erector spinae plane block (ESPB) is an interfacial plane block that provides truncal analgesia. Originally described in 2016 as an analgesic technique for thoracic neuropathic pain, ESPB has since been applied in abdominal procedures. While the mechanism of ESBP requires further investigation, some postulate the target to be the ventral rami of spinal nerves. Recent randomized trials have showed ESPB to reduce pain scores in cardiac and breast surgeries.

Since Blanco et al. first described the Quadratratus lumborum block (QLB) in 2007, its use in abdominal surgeries has been shown to be superior to the transversus abdominis plane (TAP) block for postoperative analgesia in this group of patients. Dam et al. defined the transmuscular approach (QL-TM) for this block.

Regarding major lower abdominal surgery, epidural analgesia was shown to be the gold standard time-tested technique for providing postoperative analgesia, but due to its possible complications, contraindications, there is a need for other equally efficient analgesic techniques.

Study Design:

This is a prospective randomized clinical trial. The patients will be randomly assigned into three equal comparable groups, each of them contains 30 patients, using computer-generated random numbers.

Each patient signed an informed consent form for block interventions and participation in the study. Patients 'age between 18 and 65 years with American Society of anesthesiology (ASA) physical status II-III-IV, who will be scheduled for an elective open total abdominal hysterectomy will be included in the study. Ultrasound guided nerve blocks and epidural injection will be applied after induction of general anesthesia.

The first group will receive bilateral Ultrasound guided erector spinae plane (ESP) block which is a relatively new block technique and many case reports show the efficacy of this technique for different uses. To perform ESP block in the lateral position bilaterally ,the skin will be disinfected with 70% alcohol bilaterally and a linear transducer is placed in a longitudinal parasagittal orientation and erector spinae muscle, trapezius muscle, rhomboid major muscle (rhomboid major muscle is absent below T6 level) and transverse process are visualized and local anesthetic is injected (0.25% bupivacaine 20 ml in each side) in the area between transverse process and erector spinae muscle at T10 level [19]. Hadi Ufuk Yِrükoğlu et al have been using this technique in their clinic for many different indications and the results are promising.

The second group of patients will receive quadratus lumborum block which will be done in the lateral decubitus position. Right block will be performed; the patient will then repositioned for the left block. An ultrasound device will be used, in which a convex probe with broadband (5-8 MHz) will be placed in the mid-axillary line just above the iliac crest to identify the three muscles of the anterior abdominal wall (transversus abdominis, internal oblique, and external oblique). Then, scan dorsally to keep the transverse orientation until seeing the aponeurosis of the transverses abdominus muscle and by following this aponeurosis, QL muscle will be visualized with its attachment to the lateral edge of the transverse process of the L2 vertebral body and visualize the thoracolumbar fascia at the lateral edge of the QL muscle. The view of the psoas major muscle anteriorly, the erector spinae muscle posteriorly, and the QL muscle adherent to the apex of the transverse process result in a well-known view of a Shamrock with three leaves (trifoliate). A spinal needle (20G) will be inserted in-plane from the anterior to posterior direction, and the tip of the needle will be advanced anterior to the QL muscle. The target site for injection is the plane between the quadratus lumborum and psoas major muscles. A test dose of 1 mL of saline will be injected for hydro visualization of the needle tip position and for confirming its correct positioning. This will be followed by injection of 0.25% bupivacaine 20 ml in each side . The dose should not exceed the safe limits (2 mg.kg of bupivacaine). Bupivacaine will be applied (on each side) between the quadratus lumborum muscle and the psoas major muscle in the interfascial plane, using the in-plane technique.

The third group of patients will receive lumbar epidural under strict aseptic precautions, lumbar epidural was performed for patients in Group III using a 16-gauge Touhy epidural needle by a median approach. The T12 - L1 or L1 - L2 interspaces was chosen for the injection.

The epidural space identified by the loss of resistance technique. The catheter was advanced 4 cm cephalad. When the aspiration test results for blood and cerebrospinal fluid were negative, a test dose of (3 mL) 2% lidocaine with 1: 200,000 adrenaline was given after the placement of the epidural catheter.

Then this will be followed by injection of 0.25% bupivacaine 15 ml as a single injection after induction of general anesthesia .

Study Methods:

Population of the study:

Patients scheduled for elective open total abdominal hysterectomy at the National Cancer Institute who meet the inclusion criteria.

Background and demographic characteristics:

90 patients ASA II-III-IV scheduled for elective open total abdominal hysterectomy under general anaesthesia.

Methodology:

Patients between 18-65 years old who scheduled for total abdominal hysterectomy will be enrolled in the study. Approval of the ethical committee and informed written consent from all patients will be issued. Patients will be given a full and detailed explanation of the intended study protocol and will be informed about the potential benefits of the development of a successful technique as well as the potential side-effects.

Study protocol Patients will be assessed the day before surgery in a preoperative visit for evaluating their medical status, laboratory investigations and for fulfilling all the above inclusion and exclusion criteria.

The patients will be instructed how to report pain by means of the visual analogue scale (VAS) score rating, in which 0 = "no pain" and 10 = "worst possible pain"[22]. All groups of the study will be premedicated with I.V 0.02 mg/kg midazolam 30 minutes preoperatively. Heart rate (HR), mean arterial blood pressure (MBP), oxygen saturation (SO2%) will be monitored before induction of anaesthesia (base line values), immediately before surgical incision and at 30 min intervals intraoperative.

Anesthesia Management:

Induction of general anaesthesia in all study groups will be performed using a regimen of IV 1 μcg/kg fentanyl and IV 2 mg /kg propofol. Tracheal intubation will be facilitated using 0.5 mg/kg IV of Atracurium. Anesthesia will be maintained with inhaled isoflurane with MAC 1.2-1.4% in oxygen enriched air (FiO 2=0.5) and top up doses of atracurium (0.1 mg/kg) IV will be administered as required. All patients will be mechanically ventilated aiming to keep end tidal carbon dioxide within the range of 30-35 mmHg. Additional bolus doses of fentanyl 0.5µg/kg will be given if the mean arterial blood pressure or heart rate rises above 20% of baseline values. The total intraoperative fentanyl consumption will be recorded in all study groups.

Ringer acetate will be infused in order to replace any fluid deficit, maintenance and losses.

Hypotension will be defined as MAP less than 60mmHg or less than 30% from baseline. Severe (i.e., MBP less than 60 mmHg) or prolonged (i.e., duration greater than or equal to 2 min) episodes of hypotension will be treated with 0.9% normal saline and/or 5mg ephedrine in incremental doses in order to maintain mean blood pressure above 70 mmHg. At the end of surgery the residual neuromuscular blockade will be reversed using neostigmine (0.05 mg/kg) and atropine (0.02 mg/kg), and extubation will be performed after complete recovery of the airway reflexes. The patients will be transferred to the post anaesthesia care unit where MAP, heart rate and VAS pain score will be noted immediately on arrival and at 4, 8, 12 and 24 h postoperatively. Rescue analgesia will be provided in the form of IV morphine 3 mg boluses if the pain score was >3. The total amount of morphine given in 24 h will be recorded in the three groups. Thereafter, the patients will be shifted to ward and will be given acetaminophen 1 g IV every 8 hours.

ELIGIBILITY:
Inclusion Criteria:

* ASA class II , III and IV
* 18yrs ≥ Age ≤ 65yrs
* Body mass index (BMI): 20-40 kg/m2
* Patient undergoing total abdominal hysterectomy under general anesthesia.

Exclusion Criteria:

* Age < 18yrs or > 65yrs
* Patient refusal
* known sensitivity or contraindication to drugs used in the study
* Contraindication to regional anesthesia e.g. local sepsis or coagulopathy
* History of psychological disorders and chronic pain

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Total postoperative opioid consumption | first 24 hours postoperatively
  Total postoperative morphine consumption till the first 24 hours postoperatively

SECONDARY OUTCOMES:
Ramsay scores | at 0, 4, 8, 12, and 24 postoperatively.
  The (1 = anxious or restless or both; 2 = cooperative, orientated, and tranquil; 3 = responding to commands; 4 = brisk response to stimulus; 5 = sluggish response to stimulus; and 6 = no response to stimulus)
Visual analogue scale VAS | 0, 4, 8, 12 and 24 postoperatively.
  VAS score 0 no pain to 10 maximum pain
Total intraoperative fentanyl consumption | intraoperative
  dose of fentanyl consumption
mean arterial blood pressure. | intraoperative and 0, 4, 8, 12 and 24 postoperatively.
  changes in mean arteria blood pressure
Postoperative nausea and vomiting | 24 hours Postoperative
  Postoperative nausea and vomiting as side effects of morphine

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - National cancer Insititute, Cairo
  - Ahmed Mohamed Soliman, Giza

IPD SHARING:
Plan to Share IPD: Undecided
till publication